CLINICAL TRIAL: NCT00005638
Title: Phase I Trial of Combined Modality Irinotecan, Cisplatin, and Concurrent Radiation Therapy for Patients With Locally Advanced Esophageal Cancer
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Esophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-081; CDR0000067794 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1766
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage II gastric cancer; stage III gastric cancer; stage II esophageal cancer; stage III esophageal cancer; adenocarcinoma of the stomach; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Cisplatin; Irinotecan; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: irinotecan hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of chemotherapy plus radiation therapy in treating patients who have advanced cancer of the esophagus.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose limiting toxicity of irinotecan when given weekly with cisplatin and concurrent external beam multifield radiotherapy in patients with locally advanced carcinoma of the esophagus or gastroesophageal junction.
* Determine the maximum tolerated dose and the recommended phase II dose of irinotecan in this regimen in this patient population.
* Evaluate the complete response rate in these patients to one course of induction chemotherapy followed by concurrent chemotherapy and radiotherapy.

OUTLINE: This is a dose escalation study of irinotecan.

Patients receive induction chemotherapy with cisplatin IV over 30 minutes followed by irinotecan IV over 30 minutes on days 1, 8, 15, and 22. Following 2 weeks of rest, patients begin chemoradiation. Patients receive cisplatin and irinotecan as above on days 1, 8, 22, and 29 and radiotherapy once daily 5 days a week for 5-6 weeks.

Cohorts of 3-6 patients receive escalating doses of irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities.

Patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma or adenocarcinoma of the esophagus or gastroesophageal junction

  * T1, N1, M0 or T2-4, Nx, M0

    * No supraclavicular or celiac lymph nodes
* Previously untreated, newly diagnosed tumors OR
* Prior resection without adjuvant therapy with local regional failure

  * Positive microscopic margin on resection of all gross disease allowed provided no metastatic disease
* No positive malignant cytology of the pleura, pericardium, or peritoneum
* No biopsy proven tumor invasion of the tracheobronchial tree or tracheoesophageal fistula

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100% OR
* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* No known Gilbert's disease

Renal:

* Creatinine no greater than 1.5 mg/dL
* No hypercalcemia

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* No myocardial infarction within the past 6 months
* No uncontrolled hypertension

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other severe concurrent conditions (e.g., severe uncontrolled diabetes, uncontrolled infections, or cerebral vascular disease)
* No other malignancy within the past 5 years except basal cell carcinoma of the skin or carcinoma in situ of the cervix
* No history of seizure disorder currently receiving phenytoin, phenobarbital, or other antiepileptic medication
* No other concurrent medical or psychiatric condition or disease that would preclude study entry

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for esophageal cancer including adjuvant chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for esophageal cancer including adjuvant radiotherapy
* No prior mantle, chest, pelvic, or hemibody radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No concurrent prochlorperazine on day of irinotecan administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Ilson, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- [Result] Ilson DH, Bains M, Kelsen DP, O'Reilly E, Karpeh M, Coit D, Rusch V, Gonen M, Wilson K, Minsky BD. Phase I trial of escalating-dose irinotecan given weekly with cisplatin and concurrent radiotherapy in locally advanced esophageal cancer. J Clin Oncol. 2003 Aug 1;21(15):2926-32. doi: 10.1200/JCO.2003.02.147. PMID 12885811